CLINICAL TRIAL: NCT06740981
Title: Nutrition in Critically Ill Patients Undergoing Non-Invasive Ventilation: a Prospective Single-Center Study
Brief Title: Nutritional Intake in Patients on Noninvasive Ventilation: a Prospective Observational Study
Acronym: PRO-NUTRINIV
Status: Not yet recruiting | Type: Observational
Sponsor: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Principal Investigator, Francesca Moretto, Principal Investigator, Università degli Studi del Piemonte Orientale Amedeo Avogadro
Other Study IDs: CE309/2024
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Malnutrition or Risk of Malnutrition; Acute Respiratory Failure
Keywords: noninvasive ventilation; nutrition; critical illness
MeSH Terms: conditions — Malnutrition; Critical Illness | interventions — Diet Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Noninvasively ventilated patients: For patients admitted with acute respiratory failure requiring noninvasive ventilation, a food diary will be collected for five days.
  Interventions: Other: Food diary

INTERVENTIONS:
Other: Food diary — A food and beverage diary will be collected for five days starting from the initiation of noninvasive ventilation, with caloric and protein intake quantified by a Nutrition Physician Specialist.

SUMMARY:
The primary objective is to quantify the caloric and protein intake in adult participants with acute respiratory failure who start a noninvasive ventilation treatment. The main question is:

- Are participants meeting their caloric and protein target during noninvasive ventilation treatment? Participants will complete a five-day food diary collection starting from the initiation of noninvasive ventilation treatment.

DETAILED DESCRIPTION:
Background:

Nutrition is a fundamental component of Intensive Care Unit (ICU) therapy. Critically ill patients have an increased risk of developing malnutrition early from the ICU admission, a factor strongly associated with higher risks of complications, prolonged ICU/hospital stays, and increased ICU readmission and mortality rates. Malnutrition in critical patients occurs due to underlying acute disease, leading to elevated catabolic stress. The use of noninvasive ventilation (NIV) has significantly increased over the past twenty years, becoming a cornerstone of acute respiratory failure (ARF) treatment. Respiratory support is provided through an interface, usually a mask or a helmet, which often poses a significant obstacle to nutrition delivery, making oral intake impossible and necessitating the initiation of enteral (EN) or parenteral nutrition (PN). These methods can both increase patient discomfort due to nasogastric (NG) tube and central line positioning and management. While critical care guidelines for nutritional management of mechanically ventilated patients are well established, data and recommendations for patients on NIV are still limited. A retrospective study conducted by our team in the intensive care unit (data not yet published) revealed a malnutrition prevalence of 70% among patients undergoing NIV on the fifth day of hospitalization.

Objectives of the Study:

The primary objective of this study is to quantify the caloric and protein intake of patients undergoing noninvasive ventilation (NIV) in intensive care units, sub-intensive care units, and hospital wards. Secondary objectives are to assess the potential association between clinical characteristics, nutritional therapy features, and the failure to achieve caloric and protein intake targets, to evaluate complications associated with NIV to analyze differences between the actual caloric and protein intake and the recommended targets based on the type of respiratory failure (hypoxemic vs. hypoxemic-hypercapnic) for which NIV treatment is initiated.

Methods:

A monocentric prospective observational study to be conducted in the general intensive care unit (ICU), intermediate care unit of Emergency Medicine and Surgery (MECAU), Cardiology Intermediate Care Unit, cardiology and internal medicine wards of the University Hospital Maggiore della Carità in Novara.

The study will include adult patients admitted to the specified units who undergo NIV treatment for acute respiratory failure caused by various conditions (e.g., cardiogenic pulmonary edema, pneumonia, exacerbation of chronic obstructive pulmonary disease). All patients admitted to the hospital requiring the initiation of noninvasive ventilation (NIV) for acute respiratory failure within 24 hours of admission will be evaluated for inclusion in the study.

For all patients meeting the prespecified inclusion criteria and without exclusion criteria, the following data will be collected:

* Patient related data: demographic and biometric characteristics, i.e. age, sex, height (reported by the patient or a family member), weight, body mass index (BMI), calf circumference, and any weight loss over the last six months; admission diagnosis and the cause of acute respiratory failure requiring NIV treatment; comorbidities; NRS 2002 (Nutritional Risk Screening) score; laboratory values; documentation of any pressure ulcers present before NIV initiation.
* Food Diary: documentation of the actual composition of meals consumed (breakfast, lunch, dinner, and other), with precise quantification of food and liquid intake to create a five-day food diary, collected by nurses or healthcare workers (OSS) responsible for meal delivery, noting who selects the meal (patient or healthcare provider); reasons for any missed meals and the presence of fever (with the recorded temperature) will also be documented to define the patient's daily catabolic status. Caloric and protein intake will later be calculated based on the food diary in collaboration with the hospital's Dietetics and Clinical Nutrition Service.
* NIV Treatment: settings, interface used, hours of ventilation and other devices used during breaks or meals, complications during treatment.
* Hospitalization Data: length of hospital stay and in-hospital mortality. Data Collection Tools: clinical data will be recorded in a specific data collection form (attached) completed by the nursing, OSS, and medical staff involved in the study, while laboratory and hospitalization data will be gathered from hospital programs accessible via the University Hospital Maggiore della Carità's internal network.

Sample Size: a retrospective study conducted by our team in the intensive care unit (data not yet published) revealed a malnutrition prevalence of 70% among patients undergoing NIV on the fifth day of hospitalization. With a confidence level of 95%, a sample size of 126 subjects is required to estimate a malnutrition prevalence of 70% on the fifth day of NIV initiation with a precision of ±8%.

Statistical Analysis: descriptive statistics will be used to summarize the characteristics of the included patients, categorical variables will be presented as numbers and percentages, while continuous variables will be expressed as means (± standard deviation, SD) or medians [interquartile range, IQR]. T-test or Mann-Whitney U test will be applied for differences between means or medians of continuous variables, respectively, while Chi-square or Fisher's exact test will be used for categorical variables. For comparisons involving more than two groups analysis of variance (ANOVA) or Kruskal-Wallis test will be employed for continuous variables and Chi-square test will be used for categorical variables with multiple comparisons. A multivariable regression model will be applied to examine associations between clinical outcomes (dependent variables) and patient clinical characteristics or nutritional therapy features (independent variables). A p-value of <0.05 will be considered statistically significant for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or more
* Hospitalization in the participant ordinary wards, intermediate care units and intensive care unit at the Maggiore della Carità University Hospital, Novara, Italy
* Admission for acute respiratory failure of any cause requiring noninvasive ventilation treatment within 24 hours from hospital admission

Exclusion Criteria:

* Palliative noninvasive ventilation treatment
* Contraindication to oral nutrition from hospital admission
* Patients admitted for surgical or gastroenterological diagnosis
* Severe immunocompromised patients or patients undergoing therapies contraindicating oral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the participant wards, intermediate or intensive care units for acute respiratory failure from any cause, undergoing noninvasive ventilation within 24 hours from hospital admission and without exclusion criteria, will be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Caloric intake | Data will be collected on a daily food diary for five days from the start of noninvasive ventilation treatment
  Analysis of daily caloric intake per kilogram in patients undergoing noninvasive ventilation for acute respiratory failure
Protein intake | Data will be collected on a daily food diary for five days from the start of noninvasive ventilation treatment
  Analysis of daily protein intake per kilogram in patients undergoing noninvasive ventilation for acute respiratory failure.
Caloric and protein adequacy | Discrepancy will be analyzed daily for five days from the start of noninvasive ventilation treatment
  Analysis of the discrepancy between patients' actual caloric and protein intake and the caloric and protein target recommended in the critically ill patients guidelines.

SECONDARY OUTCOMES:
Risk factors for undernutrition | This evaluation will consider undernutrition as a dichotomous outcome during the five days of data collection
  Evaluation of potential associations between patient clinical and nutritional characteristics and undernutrition
Noninvasive ventilation complications | Complication occurrence will be evaluated during the five days of data collection
  Occurrence of noninvasive ventilation treatment-related complications
Caloric and protein adequacy | Discrepancy will be analyzed daily for five days from the start of noninvasive ventilation treatment
  Analysis of the discrepancy between patients' actual caloric and protein intake and the caloric and protein target recommended in the critically ill patients guidelines, according to the type of respiratory failure, hypoxemic vs hypoxemic-hypercapnic.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Maggiore della Carità, Novara, Novara, Italy

IPD SHARING:
Plan to Share IPD: No